CLINICAL TRIAL: NCT02060604
Title: A Randomised Controlled Trial of Ranibizumab With and Without Ketorolac Eyedrops for Exudative Age-related Macular Degeneration
Brief Title: Pilot Study of Ranibizumab With and Without Ketorolac Eyedrops for Exudative Age-related Macular Degeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Andrea Russo, MD, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSAIDs_01
Record Dates: First submitted 2014-02-08; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Wet Macular Degeneration
Keywords: ketorolac; NSAIDs; wet macular degeneration; choroidal neovascularization
MeSH Terms: conditions — Wet Macular Degeneration; Choroidal Neovascularization | interventions — Ketorolac; Ranibizumab

ARMS (2):
- Ketorolac + Ranibizumab (Experimental): 3 monthly ranibizumab, then as needed plus ketorolac eyedrops TID
  Interventions: Drug: Ketorolac + Ranibizumab
- Ranibizumab Alone (Active Comparator): 3 monthly ranibizumab, then as needed
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ketorolac + Ranibizumab — 3 monthly ranibizumab, then as needed Ketorolac TID
  Arms: Ketorolac + Ranibizumab
Drug: Ranibizumab — 3 monthly ranibizumab, then as needed
  Arms: Ranibizumab Alone

SUMMARY:
The addition of an anti-inflammatory agent could be a valid option for controlling choroidal neovascularization, as simply inhibiting VEGF addresses neither the multifactorial pathogenesis of choroidal neovascularization nor the underlying cause of VEGF production.

ELIGIBILITY:
Inclusion Criteria:

1. ability to provide written informed consent and comply with study assessments for the full duration of the study;
2. age >40 years;
3. presence of treatment-naïve neovascular AMD with a visual acuity between 20/25 and 20/200 on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. Inclusion criteria for AMD were neovascularisation, fluid, or haemorrhage under the fovea.

Exclusion Criteria:

1. any previous intravitreal treatment;
2. previous laser treatment in the study eye;
3. myopia >7 dioptres in the study eye;
4. concurrent eye disease in the study eye that could compromise visual acuity (eg, diabetic retinopathy, advanced glaucoma);
5. concurrent corneal epithelial disruption or any condition that would affect the ability of the cornea to heal;
6. known sensitivity to any component of the formulations under investigation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
mean change in study eye visual acuity as measured by the best-corrected ETDRS letter score | 12 months

SECONDARY OUTCOMES:
mean change in central macular thickness | 12 months
mean number of intravitreal injections over the 12-month period | 12 months
adverse ocular events at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Russo, MD, Principal Investigator — University of Brescia, Italy; Luisa Delcassi, MD, Study Chair — University of Brescia, Italy; Francesco Semeraro, Professor, Study Director — University of Brescia, Italy
Locations (1):
- Spedali Civili di Brescia, Brescia, BS, Italy